CLINICAL TRIAL: NCT00003566
Title: Pre-Resection Minimally Invasive Surgical Restaging of Stage III (Mediastinal Node Positive) Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Thoracoscopy in Patients With Stage IIIA Non-Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-39803; U10CA031946 (NIH); CLB-39803; CDR0000066632 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- video-thorascopy + surgery (Experimental): Patients will undergo ipsilateral video-thorascopic evaluation. Patients may undergo surgery at the discretion of the surgeon and treating physicians.
  Interventions: Procedure: videothoracoscopy

INTERVENTIONS:
Procedure: videothoracoscopy

SUMMARY:
RATIONALE: Diagnostic procedures such as thoracoscopy may help to measure a patient's response to previous treatment.

PURPOSE: Diagnostic trial to determine the accuracy of thoracoscopy in patients who have stage IIIA non-small cell lung cancer.

DETAILED DESCRIPTION:
OUTLINE: The purpose of this study is to test the usefulness and safety of restaging the patient's cancer by a procedure called a thoracoscopy. Restaging is a process by which physicians measure the response of the patient to treatment. The primary and secondary objectives are described below.

OBJECTIVES:

Primary Objective:

1. Evaluate the feasibility of using videothoracoscopy to access and identify residual viable cancer in mediastinal lymph nodes and/or evaluate for other conditions which render patients unresectable (pleural carcinomatosis or T4 primary tumors) following prior mediastinoscopy and a period of neoadjuvant therapy for Stage IIIA N2 non-small cell lung cancer.

Secondary Objectives:

1. Evaluate the safety (morbidity and mortality) of pre-resectional, thoracoscopic restaging of patients who have undergone prior mediastinoscopy and induction therapy for Stage III (N2) NSCLC.
2. Assess the accuracy (false-negative rate) of thoracoscopic mediastinal node restaging after prior mediastinoscopy and induction therapy.

ELIGIBILITY:
1. Histologic Documentation: All patients must have histologic documentation of Stage IIIA non-small cell lung cancer on the basis of involved N2 nodes from a documented mediastinoscopy performed prior to induction therapy. Previously treated relapsed patients are not eligible.
2. Prior Treatment: greater than or equal to 2 cycles of chemotherapy with or without radiotherapy (greater than or equal to 40 Gy) or radiotherapy alone (greater than or equal to 40 Gy) must be completed within 60 days of registration.
3. No distant metastatic disease or local disease progression. Patients with responding or stable local disease are eligible. Those with local disease progression defined as a 25% increase in local tumor size or the appearance of new areas of malignant disease are ineligible.
4. No previous intrapleural surgery on the ipsilateral side.
5. ECOG Performance Status: 0-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 1998-09; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jaklitsch, MD, Study Chair — Dana-Farber/Brigham and Women's Cancer Center
Locations (72):
- United States (71):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital Comprehensive Cancer Center, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Helen and Harry Gray Cancer Institute at Good Samaritan Medical Center, West Palm Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Lakeland Medical Center - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - NorthEast Oncology Associates, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
  - Ministry Medical Group - Northern Region, Rhinelander, Wisconsin
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico

REFERENCES:
- [Result] Jaklitsch MT, Gu L, Harpole DH, et al.: Prospective phase II trial of pre-resection thoracoscopic (VATS) restaging following neoadjuvant therapy for IIIA(N2) non-small cell lung cancer (NSCLC): results of CALGB 39803. [Abstract] J Clin Oncol 23 (Suppl 16): A-7065, 636s, 2005.